CLINICAL TRIAL: NCT04515771
Title: Improving Patient-provider Communication to Reduce Mental Health Disparities (CDA 16-153)
Brief Title: Improving Patient-Provider Communication to Reduce Mental Health Disparities
Acronym: PARTNER-MH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: CDX 20-003
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Healthcare Disparities; Mental Health
Keywords: Social Determinants of Health; Minority Health; Veterans Health; Patient Participation; Patient Navigation; Mental Health Services
MeSH Terms: conditions — Psychological Well-Being; Patient Participation

STUDY DESIGN:
Intervention Model Description: The study consisted of two groups, an active treatment group and a waitlist control group. Participants randomized to the active treatment group received the peer-administered intervention program for 6 months and then were followed for 3 months after completion of the program. The waitlist control group received the peer-administered intervention program for 6 months following a 6-month waiting period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active PARTNER-MH (Experimental): Participants in this arm received the intervention immediately after study enrollment. They continued to receive usual mental health services in addition to intervention.
  Interventions: Behavioral: PARTNER-MH
- Waitlist Control (Other): The waitlist control arm participants received usual mental health services. They were offered to receive the intervention after the 6-month wait period.
  Interventions: Behavioral: PARTNER-MH

INTERVENTIONS:
Behavioral: PARTNER-MH — The study intervention consisted of a 6-month, manualized, peer-led navigation program. It involved assessing and addressing patients' unmet social needs and barriers to care, delivery of peer support services, navigation to VA mental health services, and psychoeducation.

SUMMARY:
The purpose of this study was to develop and pilot test an intervention to reduce mental health disparities for racially and ethnically minoritized Veterans receiving outpatient VA mental health services. The program was delivered by trained VA peer navigators. The specific aims of the program were to enhance navigation of mental health services, increase patient engagement, and improve patient-provider communication.

Study participants were randomized into one of two study groups, which determined when they received the study intervention. Regardless of study group, participants had the opportunity to receive services in addition to their regular mental health treatment (either immediately after enrollment into the study or after a 6-month waiting period).

Participants were asked to complete study questionnaires at different timepoints throughout the study to assess their overall satisfaction with the study program and the mental health services that they received. Some participants also completed an interview to discuss their experience in the program.

ELIGIBILITY:
Inclusion Criteria:

To be eligible:

* Must be a Veteran belonging to a racial/ethnic minoritized group
* Must be actively receiving mental health care in the Outpatient Mental Health Clinic at Veteran Health Indiana (Richard L. Roudebush VA Medical Center)
* Must have started receiving mental health care as a new patient in the Outpatient Mental Health within 12 months prior to enrollment into the study

Exclusion Criteria:

Not eligible if:

* Is a Veteran not belonging to a racial/ethnic minoritized group
* Not actively receiving mental health care in the Outpatient Mental Health Clinic at Veteran Health Indiana (Richard L. Roudebush VA Medical Center)
* Started receiving mental health care as a new patient in the Outpatient Mental Health outside of the 12-month window

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johanne Eliacin, PhD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Final research datasets underlying all publications reporting results of VA research can be made available, upon FOIA request. Upon request, a limited dataset will be made available for other researchers for the purposes of validation of findings. The limited dataset will include de-identified data relevant to the specific request. Independent research groups can view relevant data to evaluate the extent that data sources support conclusions made by authors in published studies as well as observe additional emergent findings and view supplemental details that might not be included in publications.
Supporting Information: Study Protocol, CSR
Time Frame: Data will become available 6 months after publication.
Access Criteria: Upon request, the Research Service will consider requests for the final data sets underlying the publications to be provided to the public. These requests for access will be reviewed by the Richard L Roudebush VA Medical Center R&D Committee and Associate Chief of Staff (ACOS) and addressed within a reasonable timeframe. Final data may have variable formats and will be converted to a uniform format, when allowable. No PHI or VASI, if any, will be shared after publication, unless approved by the facility Privacy Officer for a FOIA request. Data sets will be de-identified and anonymized and VASI removed per FOIA. Only authorized research personnel as approved by the ACOS in agreement with the PI, will have access to the data. Data will be securely stored on a VA Research network drive behind the VA firewall. The project will have an assigned secure space for storage on the network drive to protect compartmentalized housing of data to include raw data, working data, and final data sets.

REFERENCES:
- [Derived] Eliacin J, Matthias MS, Cameron KA, Burgess DJ. Veterans' views of PARTNER-MH, a peer-led patient navigation intervention, to improve patient engagement in care and patient-clinician communication: A qualitative study. Patient Educ Couns. 2023 Sep;114:107847. doi: 10.1016/j.pec.2023.107847. Epub 2023 Jun 13. PMID 37331280
- [Derived] Eliacin J, Burgess D, Rollins AL, Patterson S, Damush T, Bair MJ, Salyers MP, Spoont M, Chinman M, Slaven JE, Matthias MS. Outcomes of a peer-led navigation program, PARTNER-MH, for racially minoritized Veterans receiving mental health services: a pilot randomized controlled trial to assess feasibility and acceptability. Transl Behav Med. 2023 Sep 12;13(9):710-721. doi: 10.1093/tbm/ibad027. PMID 37130337
- [Derived] Eliacin J, Burgess DJ, Rollins AL, Patterson S, Damush T, Bair MJ, Salyers MP, Spoont M, Slaven JE, O'Connor C, Walker K, Zou DS, Austin E, Akins J, Miller J, Chinman M, Matthias MS. Proactive, Recovery-Oriented Treatment Navigation to Engage Racially Diverse Veterans in Mental Healthcare (PARTNER-MH), a Peer-Led Patient Navigation Intervention for Racially and Ethnically Minoritized Veterans in Veterans Health Administration Mental Health Services: Protocol for a Mixed Methods Randomized Controlled Feasibility Study. JMIR Res Protoc. 2022 Sep 6;11(9):e37712. doi: 10.2196/37712. PMID 36066967

RESULTS

PARTICIPANT FLOW:
Groups:
- Active PARTNER-MH: Participants in this arm received the intervention immediately after study enrollment. They continued to receive usual mental health services in addition to intervention.
  PARTNER-MH was a 6-month, manualized intervention delivered by VA peer support specialists/navigators. The intervention involved assessing and addressing patients' barriers to care and unmet social needs. It also included navigation to VA mental health services, provision of peer support and psychoeducation to increase patients' engagement in mental health services and to improve their communication with mental health clinicians.
- Waitlist Control: During the 6-month waiting period, participants in this arm received usual mental health services. They had the option to receive the intervention after the wait period.
Period: Period 1: 6 Month Randomized Period
Arm/Group | Active PARTNER-MH | Waitlist Control
Started | 30 | 20
Completed | 18 | 18
Not Completed | 12 | 2
Not completed — Lost to Follow-up | 9 | 1
Not completed — Withdrawal by Subject | 3 | 1
Period: Period 2. 6 Month Waitlist Crossover
Arm/Group | Active PARTNER-MH | Waitlist Control
Started | 0 (No new participants were enrolled in the active arm at phase 2.) | 12 (12 participants form the waitlist control arm in phase 1 opted to receive the intervention in phase 2.)
Completed | 0 | 7
Not Completed | 0 | 5
Not completed — Lost to Follow-up | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Active PARTNER-MH: The Active PARTNER-MH arm will test the intervention program starting immediately after enrollment in the study. Participants enrolled into this arm will continue to receive normal mental health services in addition to the peer-administered intervention.
  PARTNER-MH: The study intervention consists of a peer navigation program developed by the study team. The navigation program focuses on navigating VA mental health services, as well as patient engagement in mental health services and patient-provider communication. The intervention will last for 6 months, during which the participant will commit to regularly meeting with their peer specialist (interventionist). Peer navigation sessions will be guided by the specific aims of the study program, but in a way that is tailored to the participants' specific needs.
- Waitlist Control: The Waitlist Control arm will test the intervention program after a waiting period of 6-months following enrollment into the study. During the 6-month waiting period, participants in this arm will continue to receive normal mental health services.
  PARTNER-MH: The study intervention consists of a peer navigation program developed by the study team. The navigation program focuses on navigating VA mental health services, as well as patient engagement in mental health services and patient-provider communication. The intervention will last for 6 months, during which the participant will commit to regularly meeting with their peer specialist (interventionist). Peer navigation sessions will be guided by the specific aims of the study program, but in a way that is tailored to the participants' specific needs.
- Total: Total of all reporting groups
Arm/Group | Active PARTNER-MH | Waitlist Control | Total
Number analyzed (Participants) | 30 | 20 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 20 | 48
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 22 | 9 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — The study included individuals identified as Hispanic White and Hispanic Black. A few also selected multiple options, such as multiracial and other. The total number therefore does not add up to 100%.
  Participants
    White (Hispanic) | 3 | 0 | 3
    Black | 20 | 15 | 35
    Asian | 0 | 1 | 1
    Other | 2 | 3 | 5
    Multiracial | 5 | 1 | 6
    Hispanic | 4 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 20 | 50
Altarum Consumer Engagement (ACE) [Mean (Standard Deviation); unit: units on a scale] — The ACE is administered as a 5-level Likert scale. The subscale scores range from 5 to 25, and the total engagement score is computed by adding the 3 subscale scores and multiplying the sum by 4/3 to obtain a possible range score of 20 to 100. Higher scores represent higher patient engagement.
  units on a scale
    ACE Commitment subscale | 13.7 (4.7) | 13.6 (5.9) | 13.7 (5.2)
    ACE Informed Choice Subscale | 10.6 (4.8) | 10.4 (5.4) | 10.5 (5.0)
    ACE Navigation Subscale | 15.5 (4.4) | 14.8 (2.8) | 15.2 (3.8)
Patient Activation Measure (PAM-MH) [Mean (Standard Deviation); unit: units on a scale] — Measure Description: The PAM-MH is a 13-item questionnaire that measures an individual's perceived ability to manage illness and health behaviors. The questions are rated on a 4-point Likert-type scale (1= strongly disagree, 2=disagree, 3=agree, 4=strongly agree). Scores are then converted using Rasch analysis to a 100-point scale. Raw scores range from 13 to 52 and converted activation scores range from 0-100. Higher activation scores indicate higher level of patient activation.
  units on a scale | 51.5 (11.3) | 49.6 (11.8) | 51.5 (11.3)
Shared-Decision-Making-9 (SDM-Q-9) [Mean (Standard Deviation); unit: units on a scale] — The SDM-Q9 PARTNER-MH was adapted from Braddock et al.'s SDM-Q-9 informed decision-making scale. The original, validated SDM-Q-9 scale has 9 items measured on a 6-point Likert scale, ranging from 0=completely disagree to 5=completely agree. The total score is calculated by summing the scores of the nine items, range from 0 (minimum) to 45 (maximum). A higher score indicates a greater level of perceived SDM.
  units on a scale | 25.8 (9.1) | 28.3 (9.7) | 26.8 (9.4)
Communication Self-Efficacy (PEPPI-5) [Mean (Standard Deviation); unit: units on a scale] — The Perceived Efficacy in Patient-Physician Interactions Scale (PEPPI-5) is 5-item scale rated on a 10-point Likert scale ranging from 1 (not confident at all) to 10 (very confident) and the total score, which is the sum of all item ratings, range from 0 (minimum) to 50 (maximum). Higher scores indicate higher levels of self-efficacy. Subscale: not applicable.
  units on a scale | 35.2 (10.6) | 36.4 (11.4) | 35.7 (10.8)
Patient Health Questionnaire (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — Patient Health Questionnaire (PHQ-9) measures severity of depressive symptoms. It includes 9 items, ranging in scores from 0 (minimum) to 27 (maximum). Higher scores indicate more severe symptoms of depression.
  units on a scale | 14.9 (6.4) | 11.5 (6.3) | 13.6 (6.5)
UCLA 6 Item Loneliness Scale (ULS-6) [Mean (Standard Deviation); unit: units on a scale] — UCLA Loneliness Scale Short Form is a 6-item scale score on a 4-point Likert Scale, ranging from 1=never to 4= often. The scale has a total summed score ranging from 6 (minimum) to 24 (maximum), with higher scores indicate higher level of loneliness.
  units on a scale | 17.1 (4.2) | 14.8 (6.3) | 16.2 (5.2)
Working Alliance Inventory (WAI-SR) [Mean (Standard Deviation); unit: units on a scale] — Working Alliance Inventory -Short Revised (WAI-SR) evaluates key aspects of the therapeutic alliance between patients and their mental health providers. It includes 12 items rated on a 5-point Likert scale ranging from 1= seldom to 5= always. The WAI-SR has 3 subscales: The Goal, Task, and Bond subscales each have 4 items and scores ranging from 4 to 20. The total summed score ranges from 12 (minimum) to 60 (maximum). For research purposes, use of the overall mean scores of the WAI-SR rather than its subscales have been recommended. Higher scores indicate higher level of working alliance.
  units on a scale
    BOND subscale | 13.5 (5.7) | 15.1 (4.4) | 14.1 (5.2)
    Goal subscale | 12.7 (6.2) | 14.8 (4.1) | 13.5 (5.5)
    Task subscale | 11.8 (4.9) | 12.8 (4.5) | 12.2 (4.7)
    Total WAI-SR scores | 38.0 (15.4) | 42.6 (11.9) | 39.8 (14.2)
VR-12 Physical Function [Mean (Standard Deviation); unit: units on a scale. T-score] — VR-12 assesses mental and physical functioning. It uses five-point ordinal response choices and provides two scores: the Physical Component Summary Score (PCS) and the Mental Health Summary Score (MCS), ranging from 0 to 100. VR-12 scores are standardized using a T-score metric with a mean of 50 and a standard deviation of 10. The United States population average PCS and MCS are 50 points each and standard deviation is 10 points. Higher scores indicate better self-reported health. Clinically significant scores vary based on disease population.
  units on a scale. T-score | 42 (7.2) | 42 (8.8) | 42 (7.7)
VR-12 Mental Function [Mean (Standard Deviation); unit: units on a scale. T-score] — VR-12 assesses mental and physical functioning. It uses five-point ordinal response choices and provides two scores: the Physical Component Summary Score (PCS) and the Mental Health Summary Score (MCS), ranging from 0 to 100. VR-12 scores are standardized using a T-score metric with a mean of 50 and a standard deviation of 10. The United States population average PCS and MCS are 50 points each and standard deviation is 10 points. Higher scores indicate better self-reported health. Clinically significant scores vary based on disease population.
  units on a scale. T-score | 31 (9.2) | 35 (5.8) | 32 (8.2)
Perceived Discrimination in Healthcare Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Respondents are asked to rate their experiences on a 5-point Likert-type scale, with answers ranging from 0 (never) to 4 (always). Higher mean scores indicate more frequent experiences of discrimination in healthcare.
  units on a scale | 1.1 (0.8) | 0.9 (0.8) | 1.0 (0.8)
CollaboRATE [Mean (Standard Deviation); unit: units on a scale] — CollaboRATE consists of 3 questions, each on a scale of 0 (No effort was made) to 9 (Every effort was made). Summed scores were multiplied by 3.7037 to change the range from 0 -27 to a possible summed, continuous score range of 0 (minimum) to 100 (maximum). Higher scores represent more shared decision-making. No subscale.
  units on a scale | 73.5 (28.3) | 81.0 (26.0) | 76.5 (27.4)
Lubben Social Network Scale LSNS-6 [Mean (Standard Deviation); unit: units on a scale] — The Lubben Social Network Scale (LSNS-6) is a self-report measure consisting of 6 items, rated on a 6-point Likert scale ranging 0 to 5. The total score is the sum of all 6 items ranging from 0 to 30. A score of 12 indicates at risk for social isolation and scores less than 12 indicate social isolation. Population: This measure was added later in the study as an exploratory measure.
  units on a scale
    number analyzed (Participants) | 6 | 3 | 9
    (all) | 14.2 (7.1) | 15.7 (0.6) | 14.7 (5.7)
Consumer Assessment of Health Care Providers and Systems [Mean (Standard Deviation); unit: units on a scale. Average score.] — 5 domains all rated from 1=Never to 4= Always and total scores for each domain are summed. Domain 1: Getting timely appointments, care, and information has 3 items, with a possible score of 3 to 12. Domain 2: How well providers communicate with patients has 4 items and possible score of 4 to 16. Domain 3: Providers' use of information has 3 items, with a possible score of 3 to 12. Domain 4: Helpful, Courteous, and Respectful Staff has 2 items, with a possible score of 2 to 8. Domain 5: Patients' rating of providers has one item, rated on a scale of 0-10. Higher values indicate better outcomes
  units on a scale. Average score.
    Domain 1 | 8.8 (2.9) | 8.8 (3.0) | 8.8 (2.9)
    Domain 2 | 14.4 (2.1) | 12.9 (2.7) | 13.8 (2.4)
    Domain 3 | 9.6 (2.5) | 9.2 (2.4) | 9.4 (2.4)
    Domain 4 | 7.3 (1.0) | 7.4 (1.2) | 7.3 (1.0)
    Domain 5 | 8.4 (1.8) | 7.2 (2.3) | 7.9 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Patient Activation Measure- Mental Health (PAM-MH)
Description: Measure Description: The PAM-MH is a 13-item questionnaire that measures an individual's perceived ability to manage illness and health behaviors. The questions are rated on a 4-point Likert-type scale (1= strongly disagree, 2=disagree, 3=agree, 4=strongly agree). Scores are then converted using Rasch analysis to a 100-point scale. Raw scores range from 13 to 52 and converted activation scores range from 0-100. Higher activation scores indicate higher level of patient activation.
Time Frame: Change from Baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Waitlist Control: During the 6-month wait period, participants in this arm received usual mental health services. They had the option to receive the intervention after the wait period.
Arm/Group | Active PARTNER-MH | Waitlist Control
Number analyzed (Participants) | 18 | 18
score on a scale | 5.7 (16.5) | 9.1 (11.7)

2. Primary Outcome: Altarum Consumer Engagement (ACE) Change
Description: The ACE is administered as a 5-level Likert scale. The subscale scores range from 5 to 25, and the total engagement score is computed by adding the 3 subscale scores and multiplying the sum by 4/3 to obtain a possible range score of 20 to 100. Higher scores represent higher patient engagement.
Time Frame: Change from Baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active PARTNER-MH | Waitlist Control
Number analyzed (Participants) | 18 | 18
score on a scale | 5.5 (11.5) | 2.9 (10.4)

3. Primary Outcome: SDM-Q9 PARTNER-MH
Description: The SDM-Q9 PARTNER-MH was adapted from Braddock et al.'s SDM-Q-9 informed decision-making scale. The original, validated scale, the SDM-Q-9, has 9 items measured on a 6-point Likert Scale, ranging from 0=completely disagree to 5=completely agree. The total score is calculated by summing the scores of the nine items, range from 0 to 45. A higher score indicates a greater level of perceived SDM.
Time Frame: Change from Baseline to 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active PARTNER-MH | Waitlist Control
Number analyzed (Participants) | 18 | 18
units on a scale | 1.9 (13.5) | 1.3 (7.1)

4. Primary Outcome: Peer Coaching Experience Satisfaction Questionnaire
Description: Peer Coaching Experience Satisfaction Questionnaire is designed to collect feedback on a respondent's overall experience with a peer coach at the end of a 6-month period. Only participants in active PARTNER-MH were administered this questionnaire. This questionnaire was developed for the study. Question 1: Overall, how satisfied are you with PARTNER-MH program? Question 2: How satisfied are you with your assigned peer. Answers are rated on a Likert scale ranging from 1 (very satisfied) to 5 (very dissatisfied).
Time Frame: Administered after completion of the study program (6 months for Active PARTNER-MH )
Population: Only 14 participants answered the question.
Measure: Number; unit: participants
Arm/Group | Active PARTNER-MH
Number analyzed (Participants) | 14
participants
  Question 1 Very satisified | 6
  Question 1 Satisified | 4
  Question 1 Neutral | 2
  Question 1 Dissatisfied | 1
  Question 1 Very dissatisfied | 1
  Question 2 Very satisfied | 11
  Question 2 Satisfied | 1
  Question 2 Neutral | 1
  Question 2 Dissatisfied | 1
  Question 2 Very dissatisfied | 0

5. Primary Outcome: Trust and Satisfaction Survey Responses Change
Description: The Trust and Satisfaction Survey is a 5-item scale which assess a respondent's degree of trust toward the VA, VA mental health care services, and the study program. Respondents are asked to rate how much they agree with each of the 5 items. Items are rated on a scale ranging from 1 (strongly disagree) to 5 (strongly agree). The survey yields final scores ranging from 5 (minimum) to 25 (maximum) with higher scores representing greater trust and satisfaction. No subscale.
Time Frame: Change from Baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active PARTNER-MH | Waitlist Control
Number analyzed (Participants) | 18 | 18
score on a scale
  Trust the VA | 0.05 (0.85) | -0.13 (0.83)
  Trust the Mental Health Clinic | 0.03 (0.69) | -0.03 (0.65)
  Would recommend MH clinic | 0.16 (0.87) | -0.19 (0.64)
  Satisfied with the care I received at MH clinic | 0.24 (0.72) | -0.53 (0.72)

6. Secondary Outcome: Veteran's RAND 12-item Health Survey (VR-12) Change
Description: The Veterans Rand 12-item Health Survey (VR-12) is a 12-item scale that assesses Veterans' report of health-related quality of life. It measures mental and physical functioning. The VR-12 uses five-point ordinal response choices and provides two scores: the Physical Component Summary Score and the Mental Health Summary Score, ranging from 0 to 100. VR-12 scores are standardized using a T-score metric with a mean of 50 and a standard deviation of 10. The scores are compared to the population average, measured in standard deviations. The United States population average PCS and MCS are 50 points each. The United States population standard deviation is 10 points. Higher scores indicate better self-reported health. Lower VR-12 MCS scores indicate worse psychological distress/functioning. Clinically significant scores vary based on the condition or disease population.
Time Frame: Change from Baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active PARTNER-MH | Waitlist Control
Number analyzed (Participants) | 18 | 18
score on a scale
  VR-12 Physical Function | -4.4 (6.8) | -0.3 (7.8)
  VR-12 Mental Function | 8.3 (6.5) | -2.8 (6.8)

7. Secondary Outcome: Perceived Efficacy in Patient-Physician Interactions Scale (PEPPI-5) Change
Description: The Perceived Efficacy in Patient-Physician Interactions Scale (PEPPI-5) is 5-item scale rated on a 10-point Likert scale ranging from 1 (not confident at all) to 10 (very confident) and the total score, which is the sum of all item ratings, range from 0 (minimum) to 50 (maximum). Higher scores indicate higher levels of self-efficacy. There is no subscale.
Time Frame: Change from Baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active PARTNER-MH | Waitlist Control
Number analyzed (Participants) | 18 | 18
score on a scale | 6.5 (11.5) | 1.2 (10.2)

8. Secondary Outcome: Working Alliance Inventory Short-Revised (WAI-SR) Change
Description: Working Alliance Inventory -Short Revised (WAI-SR) evaluates key aspects of the therapeutic alliance between patients and their mental health providers. It includes 12 items rated on a 5-point Likert scale ranging from 1= seldom to 5= always. The WAI-SR has 3 subscales: The Goal, Task, and Bond subscales each have 4 items and scores ranging from 4 to 20. For research purposes, use of the overall mean scores of the WAI-SR rather than its subscales have been recommended. The scale total scores range from 12 (minimum) to 60 (maximum). Higher scores indicate higher level of working alliance. There is no cut off score for this scale.
Time Frame: Change from Baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active PARTNER-MH | Waitlist Control
Number analyzed (Participants) | 18 | 18
score on a scale
  BOND subscale | 0.7 (3.4) | 0.7 (3.6)
  GOAL subscale | 1.6 (5.7) | 1.6 (4.0)
  TASK Subscale | 1.4 (2.7) | 0.7 (5.5)
  Summed scores | 3.8 (9.9) | 2.9 (10.9)

9. Secondary Outcome: UCLA Loneliness Scale (ULS-6) Change
Description: The UCLA Loneliness Scale Short Form, (ULS-6), is a 6-item scale that assesses loneliness and is rated on a 4-point Likert Scale, ranging from 1=never to 4= often. The scale has a total summed score ranging from 6 (minimum) to 24 (maximum), with higher scores indicate higher level of loneliness.
Time Frame: Change from Baseline to 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active PARTNER-MH | Waitlist Control
Number analyzed (Participants) | 18 | 18
units on a scale | -0.6 (4.1) | -0.3 (3.9)

10. Secondary Outcome: Patient Health Questionnaire (PHQ-9) Change
Description: Measure Description: Patient Health Questionnaire (PHQ-9) measures severity of depressive symptoms. It includes 9 items, ranging in scores from 0 to 27. Higher scores indicate more severe symptoms of depression.
Time Frame: Change from Baseline to 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active PARTNER-MH | Waitlist Control
Number analyzed (Participants) | 18 | 18
units on a scale | -3.6 (6.7) | 0.1 (5.2)

11. Other Pre Specified Outcome: Lubben Social Network Scale-6
Description: The Lubben Social Network Scale (LSNS-6) is a self-report measure consisting of 6 items, rated on a 6-point Likert scale ranging 0 to 5. The total score is the sum of all 6 items ranging from 0 to 30. A score of 12 indicates at risk of social isolation and scores less than 12 indicate social isolation.
Time Frame: change in scores from baseline to 6 months
Population: Include changes in scores for patients from baseline to 6-months. This measure was added later as an exploratory measure. Only a few participants completed it.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active PARTNER-MH | Waitlist Control
Number analyzed (Participants) | 6 | 3
score on a scale | 6.3 (7.0) | 0.0 (2.6)

12. Other Pre Specified Outcome: Perceived Discrimination in Healthcare Responses
Description: Measure Description: Respondents are asked to rate their experiences on a 5-point Likert-type scale, with answers ranging from 0 (never) to 4 (always). Higher scores indicate more frequent experiences of discrimination in healthcare.
Time Frame: Change in score from baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active PARTNER-MH | Waitlist Control
Number analyzed (Participants) | 18 | 18
score on a scale | -1.9 (5.3) | -1.6 (4.5)

13. Post Hoc Outcome: CollaboRATE
Description: CollaboRATE consists of 3-items, each scored on a scale of 0-9. Scores range from 0-100. Higher scores indicate more shared decision.
Time Frame: Change in score from baseline to 6-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active PARTNER-MH | Waitlist Control
Number analyzed (Participants) | 18 | 18
score on a scale | 1.8 (8.8) | 0.4 (6.0)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and assessed from the time of study entry at baseline until the end of study participation at 6 months (primary endpoint), or 12 months for those who were in the waitlist control arm and opted to receive the intervention.
Arm/Group | Active PARTNER-MH | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/20
Other Adverse Events (participants affected / at risk) | 1/30 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active PARTNER-MH (N=30) | Waitlist Control (N=20)
non-serious adverse event (Psychiatric disorders) | 1 (1) | 0 (0) — 1 patient was hospitalized for attempted suicide.

LIMITATIONS AND CAVEATS:
The study had some limitations that should be considered. The study was conducted with a small sample at one VHA site. It was not powered to detect significant changes. Therefore, findings should be interpreted with caution. The retention rate in the study was also moderate and differed by study group. Future evaluation of PARTNER-MH should also examine outcomes over a longer period to assess patients' health services utilization and engagement in mental health treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT04515771/Prot_SAP_000.pdf